CLINICAL TRIAL: NCT05624112
Title: Open-label Exploratory Study to Evaluate the Effect of Dupilumab on Skin Barrier Function in Chinese Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Dupilumab Skin BArrier Function and LIpidomics STudy in Atopic Dermatitis in China
Acronym: BALISTAD-CN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS17250; U1111-1272-6687 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis; Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD patients (Experimental): AD patients aged ≥12 and ≤ 65
  Interventions: Drug: Dupilumab
- Healthy volunteers (No Intervention): Non-treatment healthy volunteers

INTERVENTIONS:
Drug: Dupilumab — Dupilumab solution in a pre-filled syringe for Subcutaneous injection
  Other Names: Dupixent
  Arms: AD patients

SUMMARY:
This is a 16-week, open label, exploratory study designed to investigate dupilumab's effect on skin barrier function as measured by transepidermal water loss (TEWL) before and after skin tape stripping. During the first 2 treatment weeks, patients will have 2 on-site visits/week, followed by one on-site visit/week up to Week 4, one on-site visit every two weeks from Week 4 to Week 8, and one on-site visit every 4 weeks up to Week 16 End of Treatment phase visit (EoT) thereafter.

A follow-up visit by phone 4 weeks after the last study assessment at Week 16 will end the study for each participant (End of Study: EoS). The maximum duration of the study per participant will be 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be between 12 to 65 years of age (inclusive), at the time of signing the informed consent.
* Male or Female. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Willing to refrain from applying any topical medication products on the target assessment areas throughout the study until the EoT visit unless necessary to alleviate intolerable symptoms.
* Willing to refrain taking showers or soaking in a bathtub with soaps and body washes within 6 hours before TEWL assessments.
* Willing to NOT apply any moisturizers to the areas of the skin that are targeted assessment areas during the entire study from Day -7 to the EoT visit.
* Willing and able to comply with all clinic visits and study-related procedures.
* Capable of understanding and giving signed informed consent/assent as will be described in the protocol, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. For adolescents ≥12 and <18 years of age a specific ICF must also be signed by the participant's legally authorized representative.

ATOPIC DERMATITIS PAIENTS ONLY:

* Patients with AD diagnosis according to Hanifin and Rajka criteria at least 1 year before screening.
* Investigator Global Assessment (IGA) score of ≥3 at screening (on the 0-4 scale).
* Patients with moderate to severe atopic dermatitis that are eligible to be treated with dupilumab according to package insert.
* Patients with AD must have active lesions on the upper limbs or lower limbs, with severity for lesion erythema or edema/papulation ≥2 at screening on the 0-3 scale of the ISS.
* Participants should have a non-lesional (normal looking) skin area 4 cm from the edge of the lesional area. If unable to identify non-lesional skin 4 cm from the lesional area, it is acceptable to identify normal looking skin as close to the lesion as possible.

HEALTHY VOLUNTEERS ONLY:

* Age and gender matched to a selected AD patient by study site. Adolescents aged 12 to 17 years will be matched by post puberty status, and adults aged 18 to 65 years will be matched by age as close as possible within 10 years of age.
* No current or prior dermatologic or systemic condition that could interfere with the assessments.

Exclusion Criteria:

* Medical conditions
* Previous treatment with dupilumab within 6 months prior to screening.
* Skin conditions other than AD that can confound assessments in the area of TEWL assessments in the opinion of the investigator (ie, skin atrophy, ichthyosis, Netherton syndrome, severe photo damage).
* Cracked, crusted, oozing, or bleeding AD lesions in the designated lesional assessment area leaving insufficient skin that is adequate for TEWL assessments.
* Ocular disorder that in the opinion of the investigator could adversely affect the individual's risk for study participation. Examples include -but are not limited to- individuals with a history of active cases of herpes keratitis; Sjogren's syndrome, keratoconjunctivitis sicca or dry eye syndrome that require daily use of supplemental lubrication; or individuals with ocular conditions that require the use of ocular corticosteroids or cyclosporine.
* Systemic AD treatment or phototherapy within 4 weeks of baseline.
* Topical AD treatment within 1 week of baseline. Face and neck may be treated with topical steroids during the washout period if approved by the investigator.
* Severe prior or concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study. Examples include, but are not limited to patients with short life expectancy, patients with uncontrolled diabetes (hemoglobin A1c ≥9%), patients with cardiovascular conditions (eg, Class III or IV cardiac failure according to the New York Heart Association classification), severe renal conditions (eg, patients on dialysis), hepato-biliary conditions (eg, Child-Pugh class B or C), neurological conditions (eg, demyelinating diseases), active major autoimmune diseases (eg, lupus, inflammatory bowel disease, rheumatoid arthritis, etc), other severe endocrinological, gastrointestinal, metabolic, pulmonary, psychiatric (known suicidal intentions),lymphatic diseases, or any illness(es) that resulted in prior or current use of chemotherapy or radiation . The specific justification for patients excluded under this criterion will be noted in study documents (chart notes, electronic case report forms [eCRF], screening logs, etc).
* History of hypersensitivity reaction to tape or adhesives. Prior/concomitant therapy
* Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known) prior to Day 1, whichever is longer.
* Treatment with live (attenuated) vaccine within 4 weeks before the baseline visit.

Prior/concurrent clinical study experience

* Current participation in another investigational clinical study. Other exclusions
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals (in conjunction with section 1.61 of the ICH-GCP Ordinance E6)
* Any specific situation during study implementation/course that may raise ethics considerations
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
* Planned or anticipated major surgical procedure during the patient's participation in this study.
* Pregnant or breast-feeding women or were planning to become pregnant or breastfeed during the subject's participation in this study.
* Women unwilling to use adequate birth control, if of reproductive potential and sexually active.
* Healthy volunteers with a personal history of an atopic condition.
* Healthy volunteers with use of any topical treatment anywhere except Cetaphil, Vanicream, or the preferred moisturizer not containing additives on non-targeted skin areas.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in TEWL after 5 skin tape stripping (STS) assessed on lesional skin at Week16 in AD patients. | From baseline to week16

SECONDARY OUTCOMES:
Change from baseline in TEWL before and after 10, 15 and 20 STS respectively assessed on lesional skin at Week16 in AD patients | From baseline to week16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Dermatology Hospital of Southern Medical University (Guangdong Provincial Dermatology Hospital), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS17250 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25297&tenant=MT_SNY_9011